CLINICAL TRIAL: NCT05857761
Title: Post-traumatic Headache: Phenotyping and Exploring Pathophysiological Insights and Novel Treatment Strategies
Brief Title: GAIN Symptoms: Post-traumatic Headache
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Hammel Neurorehabilitation Centre and University Research Clinic (Other); Central Denmark Region (Other)
Responsible Party: Principal Investigator, Charlotte Nygaard, Medical Doctor, PhD student, Regionshospitalet Hammel Neurocenter
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GAIN: Post-traumatic Headache
Record Dates: First submitted 2023-03-24; First posted 2023-05-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Post-Traumatic Headache; Concussion, Mild; MTBI - Mild Traumatic Brain Injury
Keywords: Post-traumatic headache; Concussion; Mild Traumatic Brain Injury
MeSH Terms: conditions — Post-Traumatic Headache; Brain Concussion

STUDY DESIGN:
Intervention Model Description: The intervention study will be conducted as a randomized, sham-controlled, parallel group clinical trial consisting of an active (n=31) and a sham group (n=31).
Who Masked: Participant
Masking Description: A computer will randomize participants to either participate in the active- or the sham group. At end of treatment participants will be asked to answer if they have received sham- or active treatment in order to assess the success of participant-blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham group (Sham Comparator): participants (n=31) will receive sham rTMS.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation (rTMS)
- Active rTMS treatment (Active Comparator): Participants (n=31) will receive active rTMS treatment.
  Interventions: Device: Active repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation (rTMS) — Five sessions of active rTMS therapy will be distributed over 2 weeks (20 Hz, 2000 pulses, 90% resting motor threshold) will be delivered to left dorsolateral pre-frontal cortex (DLPFC) around 6 months post-trauma.
  Arms: Active rTMS treatment
Device: Sham repetitive transcranial magnetic stimulation (rTMS) — Five sessions of sham rTMS therapy will be distributed over 2 weeks
  Arms: Sham group

SUMMARY:
The overall aim of the study is to advance the knowledge on the characterization and underlying pathophysiological mechanisms of persistent post-traumatic headache (PTH) with a direct impact on the ability to diagnose and manage PTH effectively. The investigators also aim to evaluate the efficacy of repetitive transcranial magnetic stimulation (rTMS), a novel intervention on PTH.

DETAILED DESCRIPTION:
Post-traumatic headache (PTH) is one of the most common and persistent symptoms following mild traumatic brain injury (mTBI), with an estimation of 18-22% developing persistent (> 3 months) PTH. PTH is highly disabling. Unfortunately, its typical characteristics and pathophysiology are poorly understood leading to its complicated and diverse management.

There is no agreement on the clinical presentation of PTH.This is largely due to the scarcity of longitudinal prospective data on large cohorts of PTH. Describing headache phenotypes longitudinally might improve disease characterization, facilitate better classification and provide evidence based-criteria of diagnosing PTH. Furthermore, exploring biomarkers associated with mTBI may provide new knowledge on the poorly understood pathophysiology of post commotional symptoms (PCS) and PTH. Additionally, there are indications of somatosensory disturbances and impaired endogenous analgesic systems in PTH patients. Assessment of somatosensory signs and symptoms in relation to pain complaints and functioning of endogenous analgesic system may also aid in better understanding of pain mechanisms in these patients. Functioning of endogenous analgesic system can be assessed using conditioned pain modulation (CPM) paradigms. Further, a curious observation in concussion patients with face and/or head pain is that they perceive painful/affected area (head and/or face region) as "swollen" or "different" without any clinical signs or obvious physical differences. Hence, such "illusions" represent body image distortions or perceptual distortion (PD) of the head or face region, and may contribute to the chronification of pain. PD can significantly affect psychosocial well-being of patients as the face/head region is a key feature of one´s identity. Unfortunately, such a distressing phenomenon has not been investigated before in these patients. Currently, no strong evidence-based treatment guidelines for PTH exist. Neuromodulation using repetitive transcranial magnetic stimulation (rTMS) targeting involved brain regions and functional networks has recently been employed to treat several chronic pain conditions including migraine. Thus, rTMS could offer an optimal new treatment strategy for PTH, as there is an evidence of brain network dysfunction in these patients.

The overall aim is to advance the knowledge on the characterization and underlying pathophysiological mechanisms of persistent PTH. The aim is also to measure the prevalence of perceived size changes (PD) of head and/or face region in patients with mild traumatic brain injury and its association with pain/PTH and other post commotional symptoms (PCS). The investigators will also evaluate the efficacy of rTMS on PTH. Deep phenotyping of PTH will be performed. Blood samples from mTBI patients will be examined for the biomarkers of PCS and PTH and the association between the biomarkers and the symptom levels of PCS, in particular PTH frequency and intensity will be evaluated. Baseline biomarker levels in the blood samples from patients with mTBI will be compared to biomarker levels in blood samples from anonymous healthy age- and sex matched controls (blood donors) or published reference intervals from the litterature. Additionally, the association between somatosensory function including CPM and the PTH frequency and intensity will be examined. Further, the effect of rTMS on headache severity and frequency (primary outcome) and somatosensory function, PD and other PCS (secondary outcome) after 1 and 3 months of stimulation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. mTBI within the last 2 to 4 months according to the diagnostic criteria recommended by the WHO task force
2. age ≥ 18 years at the time of mTBI
3. Rivermead Post-Concussion Symptoms Questionnaire (RPQ) score ≥ 3 (moderate or severe problem) for subitem headache and a diagnosis of persistent PTH attributed to mTBI according to ICHD-3.

Additionally, for study 2 and 3, subjects have to be stable on preventative headache medication. However, subjects are permitted to take ''as needed'' (PRN) medications throughout the study with documentation in a daily headache diary.

Exclusion Criteria:

1. objective neurological findings and/or acute trauma CT scan indicating neurological disease or brain damage
2. previous mTBI within the last 2 years years leading to PCS lasting ≥ 3 months. Additionally, for study 2 and 3,
3. Pre-trauma headache frequency ≥ 10 days in average per month the last 3 months prior to mTBI.
4. past history of TMS therapy or TMS-related contraindications (pacemaker, epilepsy etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of headache days of moderate to severe intensity | Prior to intervention compared to 1 month after end of treatment.
  Change in the number of headache days of moderate to severe intensity from baseline to 1-month post intervention based on a self-reported daily headache diary, a self-reported headache questionaire and Headache Impact test (HIT-6).
Changes in the concentration of biomarkers | Prior to rTMS intervention, immediately after rTMS intervention and 1 month after end of treatment
  Changes in the blood biomarkers (such as neurofilament light chain, calcitonin gene related peptide, pituitary adenylate cyclase-activating polypeptide, cytokines, mRNA, microRNA and circular RNA) and somatosensory function from baseline to immediately after the completion of intervention (rTMS) and 1 month post-rTMS.
A comparison at baseline of the blood biomarker concentrations in the mTBI patients compared to healthy controls | Prior to rTMS intervention
  Differences in the blood biomarkers (such as neurofilament light chain, calcitonin gene related peptide, pituitary adenylate cyclase-activating polypeptide, cytokines, mRNA, microRNA and circular RNA) at baseline.
Characterization of PTH headache phenotypes using a self-constructed headache questionaire. | 3 months after mTBI
  Characterization of PTH headache phenotypes into e.g. migraine-like or tension-type like using a self-constructed headache questionnaire.

SECONDARY OUTCOMES:
Change in the number of headache days of moderate to severe intensity | Prior to intervention compared to 3 months after end of treatment.
  Change in the number of headache days of moderate to severe intensity from baseline to 1-month post intervention based on a self-reported daily headache diary, a self-reported headache questionaire and Headache Impact test (HIT-6).
Change in severity of post-concussion symptoms covering physical, cognitive, and emotional symptoms. | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using the Rivermead Post-Concussion Symptoms Questionnaire (RPQ) [range 0-64 (worst)].
Change in the use of medication, non-pharmacological treatment and management strategies. | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using a self-constructed, self-reported questionaire
Change in health-related quality of life | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using the EuroQol-5 Domain (EQ-5D-5L) [5 items, range 0-100. 100 means the best health you can imagine]
Change in self-reported impact on participation and autonomy | Prior to intervention compared to 1 and 3 months after end of treatment.
  Will be measured using the Impact on Participation and Autonomy questionaire (IPAQ-DK). IPAQ DK consists of 32 items which can be answered from 0-4. Higher score corresponds to less participation and autonomy.
Change in Psychological Distress | Prior to intervention compared to 1 and 3 months after end of treatment.
  Will be measured using the Screening for Anxiety and depression (SCL-13). SCL-13 consists of 13 items from the Symptom Check List-90. Each item can be ranged from 0-4 (not at all- very much). A high score corresponds to a high level of depressive and/or anxiety symptoms.
Change in illness perception | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using the The Brief Illness Perception Questionnaire (B-IPQ). B-IPQ consists of 9 items. Each item is rated on a 0-10 scale, with higher scores indicating a more threatening perception of the illness. The total score is calculated by summing the scores of all eight items, with a possible range of 0-80. Higher scores indicate worse illness perception.
Change in Pain Catastrophizing | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using the Pain Catastrophizing Scale (PCS-DK). Consists of 13 items. Each item is ranged from 0-4. A high score corresponds to a high degree of pain catastrophizing.
Change in facial perception | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using a self-constructed, self-reported questionaire
Change in self-reported efficacy of treatment | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using Patients Global Impression of Change (PGIC-DK). 1 item ranged 0-6. A high score corresponds to a subjective improvement.
Change in how neck pain affects daily life | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using the Neck Pain Disability Index (NDI-DK). 8 items ranged 0-6. A high score corresponds to a high impact on daily life.
Changes in sleep quality | Prior to intervention compared to 1 and 3 months after end of treatment
  Will be measured using the Pittsburgh Sleep Quality Index (PSQI-DK). seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Changes in the somatosensory function. | prior to rTMS intervention, immediately after rTMS intervention and 1 month after end of treatment
  Change in the somatosensory function from baseline to immediately after the completion of intervention (rTMS) and 1 month post-rTMS.
Characterization of PTH headache phenotypes using the Headache Impact Scale. | 3 months after mTBI
  Characterization of PTH headache phenotypes into e.g. migraine-like or tension-type like using the Headache Impact Scale (HIT-6). HIT-6 is a 6 item scale. Each item is ranged from 0-5 ("never-always"). A high total score corresponds to a high impact of the headache on daily functioning.
Changes in headache phenotype using a self-constructed headache questionaire. | 3, 9 and 12 months after mTBI
  Describing changes in the headache phenotype (e.g. migraine-like or tension-type like) longitudinally using a self-constructed headache questionnaire.
Changes in headache phenotype using the Headache Impact Scale . | 3, 9 and 12 months after mTBI
  Describing changes in the headache phenotype (e.g. migraine-like or tension-type like) longitudinally using the Headache Impact Scale (HIT-6). HIT-6 is a 6 item scale. Each item is ranged from 0-5 ("never-always"). A high total score corresponds to a high impact of the headache on daily functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Feldbæk Nielsen, Proffessor, Study Director — Research Unit Hammel Neurocenter
Locations (1):
- Reseach Unit Hammel Neurocenter, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebener M, Hasselhorn HM. Validation of Short Measures of Work Ability for Research and Employee Surveys. Int J Environ Res Public Health. 2019 Sep 12;16(18):3386. doi: 10.3390/ijerph16183386. PMID 31547466
- [Background] Mollica A, Safavifar F, Fralick M, Giacobbe P, Lipsman N, Burke MJ. Transcranial Magnetic Stimulation for the Treatment of Concussion: A Systematic Review. Neuromodulation. 2021 Jul;24(5):803-812. doi: 10.1111/ner.13319. Epub 2020 Nov 12. PMID 33184973